CLINICAL TRIAL: NCT04824872
Title: A Double-Blind, Placebo-Controlled, Cross-over Trial, Evaluating Efficacy and Safety of Dasiglucagon for Treatment of Post-bariatric Hypoglycemia in Roux-en-Y Gastric Bypass (RYGB) Operated Adults
Brief Title: Efficacy and Safety of Dasiglucagon for Treatment of Post-bariatric Hypoglycemia in Roux-en-Y Gastric Bypass (RYGB) Operated Adults
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Never started
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZP4207-20123
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Hypoglycemia; Glucose Metabolism Disorders
MeSH Terms: conditions — Hypoglycemia; Glucose Metabolism Disorders | interventions — dasiglucagon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Sequence 1 (Experimental): Dasiglucagon high dose, followed by placebo, followed by dasiglucagon low dose
  Interventions: Drug: Dasiglucagon; Drug: Placebo
- Sequence 2 (Experimental): Dasiglucagn low dose, followed by dasiglucagon high dose, followed by placebo
  Interventions: Drug: Dasiglucagon; Drug: Placebo
- Sequence 3 (Experimental): Placebo, followed by dasiglucagon low dose, followed by dasiglucagon high dose
  Interventions: Drug: Dasiglucagon; Drug: Placebo
- Sequence 4 (Experimental): Dasiglucagon high dose, followed by dasiglucagon low dose, followed by placebo
  Interventions: Drug: Dasiglucagon; Drug: Placebo
- Sequence 5 (Experimental): Placebo, followed by dasiglucagon high dose, followed by dasiglucagn low dose
  Interventions: Drug: Dasiglucagon; Drug: Placebo
- Sequence 6 (Experimental): Dasiglucagon low dose, followed by placebo, followed by dasiglucagon high dose
  Interventions: Drug: Dasiglucagon; Drug: Placebo

INTERVENTIONS:
Drug: Dasiglucagon — dasiglucagon SC, low dose
Drug: Dasiglucagon — dasiglucagon SC, high dose
Drug: Placebo — placebo for dasiglucagon

SUMMARY:
The objective of the trial is to assess the effect of single subcutaneous doses of dasiglucagon versus placebo on post-prandial plasma glucose nadir following a Mixed Meal Test in Roux-en-Y Gastric Bypass (RYGB) subjects

ELIGIBILITY:
Inclusion Criteria:

* Previously undergone Roux-en-Y gastric bypass (RYGB) surgery at least 6 months prior to screening
* Previous diagnosis of post-bariatric hypoglycemia (PBH), requiring intake of oral carbohydrates.
* Body mass index (BMI) ≤ 40 kg/m2
* Fasting plasma glucose between 72-106 mg/dL (4.0-6.0 mmol/l)

Exclusion Criteria:

* History of hypersensitivity reactions to glucagon or dasiglucagon or any of the excipients
* History of insulinoma, pheochromocytoma, MEN 2A, MEN 2B, neurofibromatosis, or von Hippel-Lindau disease.
* Estimated Glomerular Filtration Rate (eGFR) < 30 mL/min/1.73 m2 or end-stage renal disease at screening
* Hepatic disease, including serum alanine aminotransferase or aspartate aminotransferase ≥ 2.5 times the upper limit of normal (ULN)
* Active malignancy, except for basal or squamous cell skin cancers
* History of a cerebrovascular accident within 6 months prior to screening
* History of myocardial infarction, unstable angina, or revascularization within 6 months prior to screening.
* Congestive heart failure, New York Heart Association Class III or IV
* Concurrent administration of β-blocker therapy
* Clinically significant ECG abnormalities at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Nadir plasma glucose concentration | From trial drug administration to 240 minutes after initiation of Mixed Meal Test

SECONDARY OUTCOMES:
Percent time spent in hypoglycemia | From trial drug administration to 240 minutes after initiation of Mixed Meal Test
  Defined as time with a plasma glucose value of 70 mg/dL (3.9 mmol/L) or less
Percent time spent in clinical significant hypoglycemia | From trial drug administration to 240 minutes after initiation of Mixed Meal Test
  Defined as time with a plasma glucose value of 54 mg/dL (3.0 mmol/L) or less
Percent time spent in target range | From trial drug administration to 240 minutes after initiation of Mixed Meal Test
  Defined as time with a plasma glucose value of 70-180 mg/dL (3.9-10.0 mmol/L)
Percent time spent in hyperglycemia | From trial drug administration to 240 minutes after initiation of Mixed Meal Test
  Defined as time with a plasma glucose value >180 mg/dL (>10 mmol/l)